CLINICAL TRIAL: NCT01680627
Title: The Effect of Computerized Alcohol Screening and Brief Intervention (CASI) on Alcohol Consumption in Adolescent Patients in the Emergency Department
Acronym: CASI
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Shahram Lotfipour, Principal Investigator, University of California, Irvine
Other Study IDs: 2011-8442
Record Dates: First submitted 2012-09-04; First posted 2012-09-07 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Alcohol Consumption
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- ADOLESCENT
  Interventions: Behavioral: CASI

INTERVENTIONS:
Behavioral: CASI

SUMMARY:
The purpose of this research is to examine the effectiveness of the Computerized Alcohol Screening and Brief Intervention (CASI) in adolescent patients in the Emergency Department at the UC Irvine Medical Center. This research study will evaluate the effectiveness of the brief intervention compared to standard of care (no intervention). Brief interventions have a high potential impact in ED. Computerized alcohol screening and brief intervention (CASI) is a fast and easy to use tool for patients and healthcare providers. CASI provides the Alcohol Use Disorders Identification Test (AUDIT-C)4, from the World Health Organization and CRAFFT3, followed by a brief intervention and customized alcohol intake recommendations for the patient. This study will also determine the effectiveness of the brief intervention in reducing alcohol use/abuse in adolescents between 12-17 years of age.

The overall goal of this study is to identify at risk alcohol use/abuse in adolescents and provide an intervention at an early stage. The current data to support alcohol and screening and brief intervention in adolescents is limited. The researchers hope that this research study will add to the overall body of knowledge in support of using the emergency department as a tool in public health, as it relates to the individual patients morbidity and mortality (pancreatitis, cirrhosis) and to the societal costs of alcohol use (lost days of work, motor vehicle collisions).

ELIGIBILITY:
Inclusion Criteria:

- Ages 12-17

Exclusion Criteria:

- Intoxicated

Ages: 12 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: EMERGENCY DEPARTMENT
Sampling Method: Non-Probability Sample
Enrollment: 235 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-06-01 (Actual); Study Completion 2015-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Irvine Medical Center, Orange, California, United States

REFERENCES:
- See also: Center for Trauma and Injury Prevention Research — http://www.ctipr.uci.edu/